CLINICAL TRIAL: NCT02094001
Title: Evaluation of Right Ventricular Function and Metabolism Following Riociguat for the Treatment of Chronic Thromboembolic Pulmonary Hypertension- Images of Rio
Brief Title: Pilot Study to Evaluate Right Ventricular Function With Riociguat in CTEPH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Lisa Mielniczuk, Medical Director, Pulmonary Hypertension Clinic, Ottawa Heart Institute Research Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20130903-01H
Record Dates: First submitted 2014-03-17; First posted 2014-03-21 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2017-06

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Riociguat therapy (Experimental): After an overnight fast, patients will undergo a 20 minute dynamic PET scan with injection of 3 MBq/kg of N-13 ammonia (NH3) to measure myocardial perfusion. Followed by a 60 min dynamic PET scan with injection of 3MBq/kg of F-18-FDG to measure glucose uptake.
  Interventions: Radiation: Cardiac PET imaging using F-18-FDG, N-13 ammonia( NH3)

INTERVENTIONS:
Radiation: Cardiac PET imaging using F-18-FDG, N-13 ammonia( NH3) — After an overnight fast, patients will undergo a 20 minute dynamic PET scan with injection of 3 MBq/kg of N-13 ammonia (NH3) to measure myocardial perfusion. Followed by a 60 min dynamic PET scan with injection of 3MBq/kg of F-18-FDG to measure glucose uptake.

SUMMARY:
Chronic thromboembolic Pulmonary hypertension(CTEPH) is characterized by obstruction of the pulmonary vasculature, leading to increased pulmonary vascular resistance, progressive pulmonary hypertension (PH) and right ventricular failure- most common cause of death for patients with PH. Riociguat, (ADEMPAS) is a member of a new class of drug recently approved in Canada for the treatment of CTEPH.

This pilot study is designed to assess if at least 24 weeks of treatment with riociguat will show changes in glucose metabolism and improved resting myocardial blood flow using positron emission tomography ( PET ) imaging to measure myocardial function. The response between both treatment naive patients as well as patients on maximally tolerated dose of riociguat with tratment duration of at least 3 months will be included.

DETAILED DESCRIPTION:
It remains unclear as to why certain patients with PH develop right heart failure. Several lines of evidence suggests alterations in right ventricular (RV) function may be precipitated by RV ischemia. This ischemia results from both decreased right coronary artery perfusion pressure and from arteriolar- capillary rarefaction. It has been proposed that this contributes to insufficient oxygen delivery needed to support the increase RV demand in right heart failure (RHF), this stimulating glycolytic shift. However, this glycolysis is insufficient to compensate for suppression of glucose oxidation in severe right ventricular hypertrophy (RVH), resulting in a state of RV hibernation and progressive RHF.

This study is designed to assess if 24 weeks of treatment with riociguat will be associated with changes in glucose metabolism and improved RV blood flow using N-13-ammonia (NH3) to measure myocardial perfusion.

We will assess the response in both treatment naive patients as well as patients who have been titrated to maximally tolerated doses of riociguat with total treatment duration of at least 3 months.

The assessment of quantitative myocardial blood flow will be combined with an advanced 3 dimensional echocardiographic assessment of RV volume and function and with cardiac magnetic resonance (MR).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to provide their written informed consent to participate in the study after having received adequate previous information and prior to any study specific procedures.
* At least 18 years of age at the time of screening.
* Receiving riociguat therapy for CTEPH.
* Patients with inoperable CTEPH or persistent or recurrent PH, after undergoing pulmonary endarterectomy.
* CTEPH diagnosis will be based on either Ventilation/ Perfusion scan (V/Q), pulmonary angiography or computed tomography pulmonary angiography..
* Clinical right heart catheterization performed confirming mean pulmonary artery pressure (mPAP >25 mmHg).
* Pulmonary vascular resistance (PVR) > 300 dyne/sec/cm5

Exclusion Criteria:

* • All types of pulmonary hypertension except Dana Point Classification Group 4 (1).

  * Patients who are currently taking Phosphodiesterase type 5 (PDE-5) inhibitors, ERAs and prostanoids ≤ 3 days prior to start of riociguat treatment.
  * Pulmonary endarterectomy surgery within 3 months of screening.
  * Epicardial coronary artery disease (Ejection Fraction <40%).
  * Previous myocardial infarction within the 3 months prior to screening.
  * Severe proven or suspected coronary artery disease (CCS Angina Classification II-IV), and/or requiring nitrates.
  * Uncontrolled arterial hypertension (systolic blood pressure> 180 mmHg and/or diastolic BP> 110 mmHg.
  * Systolic blood pressure <95mmHg.
  * Resting heart rate in an awake patient <50 beats per minute (bpm) or >105 bpm.
  * History of uncontrolled atrial fibrillation within the last 3 months prior to screening.
  * Hypertrophic obstructive cardiomyopathy.
  * Clinical evidence of symptomatic atherosclerotic disease (peripheral artery disease).
  * Pregnant or breastfeeding women or women with childbearing potential not using highly effective contraception methods.
  * Renal insufficiency (glomerular filtration rate < 30 ml/min.
  * ALT or AST > times upper limit of normal( ULN) and/or severe hepatic insufficiency.
  * Contraindication to MRI imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Evidence of changes in glucose metabolism and myocardial RV blood flow in patients treated with riociguat using PET imaging. | After 24 weeks of treatment with riociguat.
  Subjects will undergo FDG (fluorodeoxyglucose, F-18)cardiac positron emission tomography studies (PET) at baseline and 24 weeks to assess regional myocardial blood flow. The assessment of regional myocardial blood flow will be combined with 3D echocardiography and magnetic resonance (MR)

SECONDARY OUTCOMES:
Evidence of improved RV function and volumes using 3D echocardiography and magnetic resonance imagining (MRI) | baseline and 24 weeks
  The assessment of will be obtained by 3D echocardiography and MRI to evaluate RV function.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Mielniczuk, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No